CLINICAL TRIAL: NCT01875354
Title: A Prospective, Randomized, Blinded, Controlled Study Investigating the Effects of a Novel Body Weight Management Program Over 90-days and Weight Maintenance at One Year.
Brief Title: A Prospective Study Investigating the Effects of a Novel Weight Management Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmanex (Industry)
Collaborators: Utah State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-PHX-01-NU-02
Record Dates: First submitted 2013-06-05; First posted 2013-06-11 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo and Low Fat Eating Plan (Placebo Comparator): Placebo Supplement A Powder Mix Days 1 - 15, (1 packet mixed in water or favorite beverage once a day) Placebo Supplement B Days 1 - 90, (1 capsule taken three times a day with a meal) Placebo Supplement C Days 1 - 90, (2 capsules taken with morning and evening meal)
  The placebo group will be instructed to consume every day, a low fat standard of care eating plan delivering approximately 1200-1500 Kcals.
  Interventions: Dietary Supplement: Placebo and Low Fat Eating Plan
- Dietary Supplements and TR90 Eating Plan (Experimental): Supplement A Powder Mix Days 1 - 15, (1 packet mixed in water or favorite beverage once a day) Supplement B Days 1 - 90, (1 capsule taken three times a day with a meal) Supplement C Days 1 - 90, (2 capsules taken with morning and evening meal)
  Experimental group will be instructed to consume every day, dietary supplements and a moderate protein eating plan delivering approximately 1200-1500 Kcals.
  Interventions: Dietary Supplement: Dietary Supplements and TR90 Eating Plan

INTERVENTIONS:
Dietary Supplement: Dietary Supplements and TR90 Eating Plan — Supplements to maintain muscle, assist in utilization of body fat, curb appetite, support positive willpower along with TR90 Eating plan. TR90 Eating Plan will consist of approximately 30 g high quality protein along with fruit, vegetables and complex carbohydrates
  Arms: Dietary Supplements and TR90 Eating Plan
Dietary Supplement: Placebo and Low Fat Eating Plan
  Arms: Placebo and Low Fat Eating Plan

SUMMARY:
The purpose of this study is to assess the safety and efficacy of a weight management program composed of dietary supplements and a reduced calorie eating program.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18-65 years of age at the time of informed consent
2. The ability to read, speak and understand the English language in order to complete the required paper informed consent, assessments and diary
3. Access to email and to a digital camera or camera phone
4. Willing and able to provide written informed consent
5. Willing and able to comply with the study restrictions, procedures and assessments and attend regularly scheduled clinic visits
6. Willing and able to accommodate being contacted by the study staff for telephone call visits, follow-up contacts, and study visit reminders
7. BMI is equal to or greater than 25 and less than or equal to 40 kg/m2
8. Use of effective method of contraception by females of childbearing potential 30-days before the screening visit and agree to continue to practice that acceptable method of contraception for the duration of her participation in the study
9. A resting normotensive blood pressure, as defined as a systolic blood pressure between 150-90 mmHg and a diastolic blood pressure of between 95-50 mmHg, at screening visit 1(A)
10. Willing to fast for at least 8 hours prior to the study procedures being performed that require fasting measurements
11. Willing and able to follow eating program and able to consume the study supplied Supplements, Placebos and shakes (which include whey and/or egg protein) on a daily basis. Subjects that are lactose intolerant will be considered ineligible
12. Only one member per household eligible to participate in the study

Exclusion Criteria:

1. A subject that has any Axis I Psychiatric disorders according to the DSM-IV criteria that would prevent the subject from being able to comply with study requirements and/or taking anti-psychotic medication
2. Diagnosed with insomnia and is chronically using prescribed or OTC insomnia medications
3. A self-reported chronic condition that may affect subject safety
4. An HbA1c of greater than or equal to 7.0%
5. Renal insufficiency as defined by a laboratory Glomerular Filtration Rate of less than 50 mL/min/1.73 m2
6. Chronically using glucocorticoid steroids
7. Currently pregnant, planning to become pregnant during the course of the study or is breastfeeding
8. Use of antihypertensive medication(s) for less than 90 days prior to screening
9. Diagnosed with any thyroid disorder or has a clinically significant out of range laboratory value (i.e. TSH, T3 Free, and/or T4 Free) value measured at screening
10. Known allergy or intolerance to any of the ingredients contained in the Novel Supplements, placebos or shakes (cow milk proteins)
11. Planned surgical procedure during the 365 day course of the study
12. Currently participating in another clinical research study or have done so within 30 days prior to the screening visit
13. Diagnosis of milk or egg intolerance
14. Participating in another weight loss program or using another weight loss product. Subjects may enroll if they are willing to stop the weight loss program they are currently on and/or washout of the product they are using. The appropriate washout will be reviewed with the investigator or medically qualified designee on a case by case basis
15. Fasting LDL-C greater than 190 mg/dL or triglycerides greater than 400 mg/dL.
16. Unwilling to discontinue consumption of green or black tea or green or black tea extracts beginning at the screening visit and after signing of the informed consent
17. Unwilling to discontinue use of over-the-counter and/or prescribed vitamin supplements except for: multivitamins, calcium, fish oil, vitamin C, vitamin D, vitamin E, zinc or iron
18. Plans to have plastic or reconstructive surgery or any other procedure that, in the opinion of the investigator, could influence body composition, at any time during the year long study
19. Unable to lay supine for at least 30 minutes
20. Cognitive impairment that would limit ability to understand or follow diet instructions and/or comply with the study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2013-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Determine the effect of a novel weight management program on body fat mass over 90 days. | Days 0 and 90
  Evaluate changes in body measurements (weight and BMI; arm, waist, hip, thigh, claf, and ankle circumferences) and body composition (fat mass, fat free mass, % body fat) by Dual Energy X-ray Absorptiometry (DEXA) scanner.

SECONDARY OUTCOMES:
Determine the safety of novel weight management program (CBC, Comp. metabolic, lipid panel, heart rate, blood pressure and adverse events) | Throughout 1 year
Evaluate changes in body measurements (weight and BMI; arm, waist, hip, thigh, claf, and ankle circumferences) and body composition (fat mass, fat free mass, % body fat) by Dual Energy X-ray Absorptiometry (DEXA) scanner. | throughout 1 year
Determine subjective measurements of hunger and appetite from standardized questionnaires (IWQOL Hunger/Appetite and overall wellbeing) | Throughout 1 year
Determine skin carotenoid (Biophotonic Scanner) measurement changes. | Throughout 1 year
  Biophotonic Scanner utilizes raman spectroscopy to determine skin carotenoid concentrations.
Evaluate the changes in metabolism and appetite hormone levels from the baseline visit to day 90. | Days 0 and 90
  Leptin, Insulin, Adiponectin, Pancreatic Polypeptide, gLP1, C-peptide, Glucagon, Resistin and HbA1c
Evaluate the changes in inflammatory markers from the baseline visit to day 90. | Days 0 and 90
  hsCRP, IL-6 and TNF Receptors 60 and 80
Evaluate the changes in gene expression from the baseline visit to day 90. | Day 0 and 90
  Full gene arrays will be made on peripheral blood mononuclear cells. The gene expression changes will be made at baseline and day 90. There will also be a comparison back to proteins (i.e. hormones and inflammatory markers).
Evaluate resting energy expenditure and substrate utilization from baseline to days 90, 180, and 365. | Days 0, 90, 80, and 365
  Resting metabolic rate (RMR)and substrate utilization (R-values to determine wheather subjects are utilizing more fats or carbohydrates to meet energy demands) will be measured by CPET Quark.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lefevre, PhD, Principal Investigator — Utah State University
Locations (1):
- Utah State University, Logan, Utah, United States